CLINICAL TRIAL: NCT03129347
Title: Pharmacokinetic Evaluation of Nalmefene Administered Intranasally to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Nalmefene-Ph1a-001
Record Dates: First submitted 2017-04-19; First posted 2017-04-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2017-11

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — nalmefene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Nalmefene (high dose) (Experimental): Nalmefene (high dose) intranasal one time during the 17 day inpatient treatment period
  Interventions: Drug: Nalmefene
- Nalmefene and Intravail (Experimental): Nalmefene (high dose) with Intravail intranasal one time during the 17 day inpatient treatment period
  Interventions: Drug: Nalmefene
- Nalmefene (low dose) (Experimental): Nalmefene (low dose) intranasal one time during the 17 day inpatient treatment period
  Interventions: Drug: Nalmefene
- Nalmefene Intramuscular (Experimental): Nalmefene intramuscular one time during the 17 day inpatient treatment period
  Interventions: Drug: Nalmefene

INTERVENTIONS:
Drug: Nalmefene — Comparing pharmacokinetics of intranasal nalmefene to intramuscular nalmefene
  Other Names: Selincro

SUMMARY:
This study will be to compare the pharmacokinetics of nalmefene administration intranasal with and without an absorption enhancer compared to an intramuscular injection.

DETAILED DESCRIPTION:
This study will be an inpatient, double-blind, randomized, crossover study involving 14 healthy volunteers. Each subject will receive 4 treatments during the 4 dosing periods.Subjects will stay in the inpatient facility for 17 days to complete the entire study and be discharged following completion of discharge procedures at the end of the last period. Subjects will be called 3 to 5 days after discharge to inquire concerning adverse events and concomitant medications since discharge. After obtaining informed consent, subject will be screened for eligibility. ON the day after clinic admission, subjects will be administered the intranasal-formulated drug in randomized order with 4 days between doses; the intramuscular dose will be administered during the fourth (last) treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 to 55 years of age
* Provide written informed consent
* Body Mass index (BMI) ranging from 18 to 32 kg/m2
* Adequate venous access
* No clinically significant concurrent medical conditions
* Males subjects must agree to use an acceptable method of birth of contraception with female partners as well as not to donate sperm throughout the study and for 90 days after the last study drug administration
* Female subjects of child bearing potential must agree to use an acceptable method of birth control from the start of screening until 30 days after completing the study. Oral contraceptives are prohibited
* Agree not to ingest alcohol, drinks containing xanthine >500 mg / day (e.g., Coca Cola, tea, coffee, etc.), or grapefruit/grapefruit juice or participate in strenuous exercise 72 hours prior to admission through the last blood draw of the study

Exclusion Criteria:

* Please contact the site for more information

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of nalmefene | 17 days
  Maximum plasma concentration, time of Maximum observed concentration and area under the concentration-time curve

SECONDARY OUTCOMES:
Safety and tolerability | 17 days
  Measure by adverse events, vital signs, ECG, clinical laboratory changes and nasal irritation following the administration of nalmefene

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kelsh, MD, Principal Investigator — Vince & Associates Clinical Research, Inc.
Locations (1):
- Vince and Associates Clinical Research, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No